CLINICAL TRIAL: NCT01420289
Title: A Randomized, Controlled Trial to Evaluate High Pressure Rapid Sequence, Intermittent Pneumatic Compression (HPIPC) for the Treatment of Intermittent Claudication, Pain and Ulcer Healing in Subjects With PAD
Brief Title: Effect of HPIPC for the Treatment of Ischemic Ulcers in Subjects With PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calvary Hospital, Bronx, NY (Other)
Responsible Party: Principal Investigator, Oscar M. Alvarez, PhD, Director, Center for Curative andPalliative Wound Care, Calvary Hospital, Bronx, NY
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-HPIPC-09
Record Dates: First submitted 2011-08-18; First posted 2011-08-19 (Estimated); Results first posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2011-08

CONDITIONS: PVD; Arterial Ulcers
Keywords: Ischemic ulcers; PAD; Intermittent Claudication Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HPIPC (Experimental): High Pressure Intermittent Pneumatic compression (HPIPC)to be performed for 45 minutes twice daily
  Interventions: Device: High pressure intermittent pneumatic compression (HPIPC)
- Excercise (Active Comparator): Walking on a graded treadmill for 45 minutes once daily
  Interventions: Behavioral: Excercise

INTERVENTIONS:
Device: High pressure intermittent pneumatic compression (HPIPC) — Apply therapy for 45 minutes twice daily
  Other Names: Bio Arterial Plus; Art Assist
  Arms: HPIPC
Behavioral: Excercise — Treadmill walking 45 minutes once daily
  Other Names: Walking on a treadmill
  Arms: Excercise

SUMMARY:
To evaluate the effects of HPIPC for the treatment of symptoms of PAD

ELIGIBILITY:
Inclusion Criteria:

* Intermittent claudication >6mo
* Ischemic ulceration or ulcer of mixed (venous) etiology
* ABI < 0.7
* Ambulatory
* Able to comply

Exclusion Criteria:

* Gangrene
* M.I. within 6mo
* Inability to walk
* Wound infection
* Systemic corticosteroids
* HBO, Apligraf, Dermagraft within 6mo
* Falsely elevated ankle to brachial index (ABI)
* Inflammatory condition affecting healing

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar M Alvarez, PhD, Principal Investigator — Director Wound Care Center
Locations (1):
- Center for Curative and Palliative wound Care, Calvary Hospital, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HPIPC: High Pressure Intermittent Pneumatic compression (HPIPC)to be performed for 1 hour twice daily
Period: Overall Study
Arm/Group | HPIPC | Excercise
Started | 18 | 16
Completed | 18 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HPIPC | Excercise | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 4 | 2 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 64 (12) | 62 (11) | 63 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 12 | 10 | 22
Region of Enrollment [Number; unit: participants]
  United States | 18 | 16 | 34

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Reduction in Wound Surface Area
Time Frame: baseline and 16 weeks
Measure: Mean (Standard Error); unit: Percent reduction in wound surface area
Arm/Group | HPIPC | Excercise
Number analyzed (Participants) | 18 | 16
Percent reduction in wound surface area | 72 (22) | 58 (15)
Statistical Analysis 1: Comparison: HPIPC vs Excercise; Test type: Superiority or Other; p = 0.086, t-test, 2 sided; Mean Difference (Final Values) = 14, 95% CI 2-sided [10 to 80], Standard Error of Mean 15

2. Secondary Outcome: Percent Improvement in Peak Walking Time
Description: Percentage Improvement in the amount of time one can walk without pain
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: Percentage Change
Arm/Group | HPIPC | Excercise
Number analyzed (Participants) | 18 | 16
Percentage Change | 96 (11) | 66 (9)
Statistical Analysis 1: Comparison: HPIPC vs Excercise; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 30, 95% CI 2-sided [10 to 100], Standard Error of Mean 11

3. Secondary Outcome: Perceived Improvement in Physical Function After 16 Weeks
Description: Percent improvement in SF-36 Quality of life (QOL) questionnaire score at baseline and at week-16.
  The higher the score on the SF-36 questionnaire the better the QOL.
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: Percent improvement in Sf-36 QOL score
Arm/Group | HPIPC | Excercise
Number analyzed (Participants) | 18 | 16
Percent improvement in Sf-36 QOL score | 70 (6) | 53 (6)

4. Secondary Outcome: Wound Pain as Determined by a Visual Analog 10 Point Scale (VAS) for Pain.
Description: Percent change (improvement)in mean VAS pain scores at baseline and at 16 weeks
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: Percent improvement in mean VAS pain sco
Arm/Group | HPIPC | Excercise
Number analyzed (Participants) | 18 | 16
Percent improvement in mean VAS pain sco | 80 (14) | 55 (9)

ADVERSE EVENTS:
Arm/Group | HPIPC | Excercise
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No